CLINICAL TRIAL: NCT02349529
Title: An Exploratory Randomised Controlled Trial of a Manualised Psychosocial Group Intervention for Young People With Epilepsy (PIE)
Brief Title: An Exploratory RCT of a Psychosocial Group Intervention for Epilepsy
Acronym: PIE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GN12KH157
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Epilepsy
Keywords: Epilepsy; psychosocial
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial group intervention (Experimental)
  Interventions: Behavioral: Psychosocial Intervention Group
- Waiting List control (Other): Participants in the waiting list control will continue in TAU but will then start the intervention once the first group of participants have completed the 3 month follow up in the psychosocial group intervention arm.
  Interventions: Other: Waiting list control

INTERVENTIONS:
Behavioral: Psychosocial Intervention Group — 6 group sessions
  Arms: Psychosocial group intervention
Other: Waiting list control — Treatment as usual
  Arms: Waiting List control

SUMMARY:
Children and young people with epilepsy are at increased risk of poorer outcomes related to emotional and psychological adjustment, peer relationship problems, lower academic attainment and mental health problems across the lifespan. Despite the well understood risks, there continues to be a lack of psychological and psychosocial support for young people with epilepsy, and a corresponding lack of evidence regarding the effectiveness of psychosocial interventions. This study aims to evaluate a manualised psychosocial group intervention for adolescents with epilepsy. A cognitive behaviour therapy approach is used, aimed at increasing awareness of how epilepsy may impact upon thoughts, feelings and activities and to develop strategies for improved psychological adjustment. In addition, an epilepsy knowledge component aimed at improving a sense of control and epilepsy self-management is included. A group delivery format allows an opportunity for social modelling, and social problem solving, helping others and relating to other young people with similar experiences. The social learning context and availability of knowledgable facilitators (an epilepsy nurse specialist and clinical psychologist) are also key aspects of the intervention. The study will allow us to establish a standard manualised group intervention that can be used throughout the UK which aims to; establish the effectiveness and desirability of this approach; improve the overall quality of life, psychological health and social integration of young people with epilepsy; and to improve epilepsy knowledge and selfmanagement skills aimed at maximising seizure control and overall management.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Diagnosis of epilepsy (controlled or refractory) of at least 6 months duration
* Between the ages of 1217 years old
* Have a reasonable level of expressive and receptive English language abilities to enable them to fully participate and contribute to the group process
* In mainstream schooling.

Exclusion Criteria:

* Formal diagnosis of Learning Disability or attendance at a school for children with Special Educational Needs
* Complex and severe mental health problems;
* Diagnosis of nonepileptic seizures in the absence of epileptic seizures
* Epilepsies occurring in the context of:

  1. Postnatally acquired structural lesions (e.g. TBI or neurooncological conditions)
  2. Immune mediated disorders (e.g. limbic or antiNMDAR encephalopathy)
  3. Metabolic disorders (e.g. GLUT1 deficiency)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the PIE group | Baseline
  Comparing participant's quality of life at baseline, completion of intervention, and at 3 and 6 month post group completion, as measured via the GEOSYP and PedsQL
Effectiveness of the PIE group | 6 weeks
Effectiveness of the PIE group | 3 months
Effectiveness of the PIE group | 6 months

SECONDARY OUTCOMES:
The Paediatric Index of Emotional Distress (PIED). | Baseline, 6 weeks, 3 months and 6 months
The Seizure Self Efficacy Scale for Children (SSEC) | Baseline, 6 weeks, 3 months and 6 months
Epilepsy Knowledge ProfileGeneral (EKPG) | Baseline, 6 weeks, 3 months and 6 months
Brief Illness Representations Questionnaire (BIPQ). | Baseline, 6 weeks, 3 months and 6 months
Participant social functioning | Baseline, 6 weeks, 3 months and 6 months
seizure control | Baseline, 6 weeks, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Liam Dorris, BSc (Hons), D.Clin.Psy, Principal Investigator — NHS Greater Glasgow and Clyde